CLINICAL TRIAL: NCT03590522
Title: Role of Amino Acids and Genetic Disorder in Pathogenesis of Heart Failure
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Reham I El-mahdy, Principal Investigator, Assiut University
Other Study IDs: Heart failure
Record Dates: First submitted 2018-07-07; First posted 2018-07-18 (Actual); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Heart Failure
Keywords: pathogenesis of heart failure; cardiac ryanodine Receptor 2; Amino acids
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group I:: Thirty heart failure patients
  Interventions: Genetic: Ryanodine Receptor 2 gene expression
- Group II:: Twenty healthy controls
  Interventions: Genetic: Ryanodine Receptor 2 gene expression

INTERVENTIONS:
Genetic: Ryanodine Receptor 2 gene expression — Ryanodine Receptor 2 gene expression will be measured by real time PCR. In addition, amino acids analysis will be measured in plasma by amino acid analyzer.

SUMMARY:
Heart failure (HF) is a continuously growing public health problem. The study aim to provide novel insights into the role of amino acids in pathogenesis of heart failure, to obtain a better understanding of cardiac ryanodine Receptor 2 role as an essential player in excitation-contraction coupling in pathogenesis of heart failure and clarify the potential value of these markers as targets for heart failure therapy

DETAILED DESCRIPTION:
Heart failure (HF) is a continuously growing public health problem. Presently, almost 40 million people are affected by heart failure worldwide. According to World Health Organization (WHO), cardiovascular diseases are number one cause of deaths globally . In developed countries, the prevalence of heart failure is approximately 1-2% of the adult population. In Egypt, the prevalence of HF with preserved ejection fraction represents about 34.2 % while heart failure with reduced ejection fraction represents 65.8 % of total heart failure cases .

A broad range of cardiac diseases, inherited disorders, and systematic diseases can result in heart failure. The situation is even more complex, as heart failure can have mixed etiologies. Heart failure itself represents a ﬁnal common pathway in response to genetic and/or environmental inﬂuences. A clear genetic identification can positively influence patient treatment and, thereby, improve prognosis. Besides, understanding the pathogenesis of genetically induced heart failure at it molecular level may lead to the development of specific individual heart failure therapies in the future.

The human heart uses large amounts of amino acids (AAs) as regulators of both myocardium protein turnover and energy metabolism, but uses few AAs as substrates for direct energy production .The heart's reliance on AAs increases during heart failure because of high myocardium anabolic activity and cardiomyocyte energy shortage. Anabolic activity of the ventricle wall is induced by both high levels of ventricular pressure and a myocardial substrate shift from fatty acid oxidation (FAOX) to glucose oxidation (GLUOX).

Various mechanisms may potentially be operating during CHF to impair arterial AAs, including inadequate protein-energy intake, body AA overconsumption, particularly in hyper metabolic states, increased remodeling activity of the heart and lung and ﬁnally, the development of pathogenic gut ﬂora. Understanding arterial AA levels could be useful to understand whether heart anabolic activity and remaining heart capacity of energy production are being threatened by low AA s and furthermore may allow us to correct altered AAs through diet and/or supplementation of speciﬁc free AAs.

A reduction in essential AAs in CHF subjects, shows the disease severity-related decline of arterial levels of those non-essential (and essential methionine) AAs with the greatest impact on myocardium energetics, anti-oxidative capacity and myocardial protein remodeling.

Calcium cycling protein and heart failure Ca2+-dependent signaling is highly regulated in cardiomyocytes and determines the force of cardiac muscle contraction. Ca2+ cycling refers to the release and reuptake of intracellular Ca2+ that drives muscle contraction and relaxation in failing hearts. Ca2+ cycling is profoundly altered, resulting in impaired contractility and fatal cardiac arrhythmias. The key defects in Ca2+ cycling occur at the level of the sarcoplasmic reticulum (SR), a Ca2+ storage organelle in muscle. Defects in the regulation of Ca2+ cycling proteins including the ryanodine receptor 2 (RyR2) a cardiac Ca2+ release channel macromolecular complexes and the sarcoplasmic/endoplasmic reticulum Ca2+ ATPase2a (SERCA2a) contribute to heart failure.

Phosphorylation of the cardiac ryanodine receptor (RyR2) phospho-site S2808 has hallmark of heart failure (HF) and a critical mediator of the physiological fight or flight response of the heart. In support of this hypothesis, mice unable to undergo phosphorylation at RyR2-S2808 (S2808A) were significantly protected against HF and displayed a blunted response to adrenergic stimulation.

ELIGIBILITY:
Inclusion Criteria:

• According to American Heart Association, patients with manifestation of heart failure (dyspnea, edema in the feet, ankles, legs or abdomen, heart palpitations) as diagnosed by clinical examination, laboratory investigations and imaging techniques.

Exclusion Criteria:

* Diabetic patients
* Neurological disorders
* Cancers.
* Obese patient
* Smokers
* Patient with chest infection

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Heart failure patients
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-01-17 (Estimated); Primary Completion 2019-03-28 (Estimated); Study Completion 2019-03-30 (Estimated)

PRIMARY OUTCOMES:
Decrease cardiac ryanodine Receptor 2 gene expression and change of amino acids levels in patients with heart failure. | Baseline
  better understanding of cardiac ryanodine Receptor 2 role as an essential player in excitation-contraction coupling in pathogenesis of heart failure and the role of amino acids in pathogenesis of heart failure

REFERENCES:
- [Background] Czepluch FS, Wollnik B, Hasenfuss G. Genetic determinants of heart failure: facts and numbers. ESC Heart Fail. 2018 Jun;5(3):211-217. doi: 10.1002/ehf2.12267. Epub 2018 Feb 19. PMID 29457878
- [Background] Bond AR, Iacobazzi D, Abdul-Ghani S, Ghorbel M, Heesom K, Wilson M, Gillett C, George SJ, Caputo M, Suleiman S, Tulloh RMR. Changes in contractile protein expression are linked to ventricular stiffness in infants with pulmonary hypertension or right ventricular hypertrophy due to congenital heart disease. Open Heart. 2018 Jan 3;5(1):e000716. doi: 10.1136/openhrt-2017-000716. eCollection 2018. PMID 29344379
- [Background] Ather S, Respress JL, Li N, Wehrens XH. Alterations in ryanodine receptors and related proteins in heart failure. Biochim Biophys Acta. 2013 Dec;1832(12):2425-31. doi: 10.1016/j.bbadis.2013.06.008. Epub 2013 Jun 14. PMID 23770282
- [Background] Alvarado FJ, Chen X, Valdivia HH. Ablation of the cardiac ryanodine receptor phospho-site Ser2808 does not alter the adrenergic response or the progression to heart failure in mice. Elimination of the genetic background as critical variable. J Mol Cell Cardiol. 2017 Feb;103:40-47. doi: 10.1016/j.yjmcc.2017.01.001. Epub 2017 Jan 6. PMID 28065668
- [Background] Aquilani R, La Rovere MT, Corbellini D, Pasini E, Verri M, Barbieri A, Condino AM, Boschi F. Plasma Amino Acid Abnormalities in Chronic Heart Failure. Mechanisms, Potential Risks and Targets in Human Myocardium Metabolism. Nutrients. 2017 Nov 15;9(11):1251. doi: 10.3390/nu9111251. PMID 29140312